CLINICAL TRIAL: NCT05050591
Title: Study for Evaluating the Clinical Effectiveness of 3D Printing for a Patient-specific Silicone Stent Airway Implant
Brief Title: Evaluating the Clinical Effectiveness of a Patient-specific Silicone Stent
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VisionAir Solutions (Industry)
Collaborators: The Cleveland Clinic (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-681
Record Dates: First submitted 2021-09-07; First posted 2021-09-20 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Prospective observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single-Arm Study (Experimental): This is a prospective trial of the clinical utility of a patient-specific silicone stent implant for patients with complex airway disease, requiring an airway stent. The aim of this study is to observe the outcomes associated with the implants. Current stents have been suboptimal for treating benign stenosis of the airway and we are seeking to create a better treatment option. We hypothesize, based on the previous compassionate-use cases, that placing a patient-specific silicone stent will effectively alleviate symptoms associated with stenosis of the airway. The main measure of effectiveness will be patient-reported outcomes.
  Interventions: Device: Patient-Specific Silicone Airway Stent

INTERVENTIONS:
Device: Patient-Specific Silicone Airway Stent — The Patient-Specific Airway Stent is a silicone stent indicated for use in adults that have stenosis of the airway. Current silicone stents have stock dimensions that do not conform to the patient's airway anatomy. The subject device takes a CT scan, thresholds out the airway from the other anatomy, and allows the physician to digitally design the stent to his/her desired dimensions. Finally, according to the physician's design, a patient-specific stent can be manufactured using additive manufacturing technology. The patient-specific stent is indicated for use with any rigid bronchoscopy/stent application system that fits the design envelope.

SUMMARY:
The goal of the trial is to establish a method, material, and patient-specific stent design that will last longer, fit better, and cause less trauma to the airway and the patient.

DETAILED DESCRIPTION:
This is a prospective trial of the clinical utility of a patient-specific silicone stent implant for patients with complex airway disease, requiring an airway stent. The aim of this study is to observe the outcomes associated with the implants. Current stents have been suboptimal for treating benign stenosis of the airway and we are seeking to create a better treatment option. We hypothesize, based on the previous compassionate-use cases, that placing a patient-specific silicone stent will effectively alleviate symptoms associated with stenosis of the airway. The main measure of effectiveness will be patient-reported outcomes.

The implant will occur on Day 0 and TDI and formal assessment for AEs will occur on Day 1.

Patients will be seen on Day 60 +/- 14 days for formal assessment including TDI and QOL, dynamic CT, and a bronchoscopy procedure will be performed as per our usual standard of care. Additional ascertainments of the TDI and QOL measurements will occur at 90 and 180 days after implantation.

A standardized assessment of the stent as well and any modification or any other treatments will be recorded. Washing for cultures will also be done per standard of care during any bronchoscopy.

ELIGIBILITY:
Inclusion Criteria: Patients will be considered for study inclusion if they have a clinical need for airway stenting defined by prior evidence of existing stents that have at least temporarily improved symptoms, but now suffer from stent complications; or those for whom a stent would be offered if an appropriate size and shape was available. Subjects must meet the following inclusion/exclusion criteria to be eligible for the study.

* Understand and voluntarily sign an informed consent form.
* Patients must be at least 22 years of age
* Patients must be able to undergo routine non-contrast CT scans of the chest
* Patient must be stable for general anesthesia and have an airway amenable to rigid bronchoscopy and stent implantation.
* The patients must have at least an expected 6 month survival.
* Patient must be able to maintain standard of care follow-up schedule and have access to standard of care medications and nebulizer machines and/or suction and oxygen as required for primary disease management.
* Patient must be able to personally provide consent and be able to describe Dyspnea and QOL and other patient-reported outcomes (PROs) required by study design
* Patient must require a stent that is within the design envelope of the patient-specific stents, as defined by COS (See Section 5.4 of this protocol for envelope)

Exclusion Criteria: Patients may be excluded if management of the airway problem can be safely and effectively treated with commercially available stents (SOC), non-stenting techniques, or surgical options.

* Patients may be excluded if the disease can be managed by simply removing prior stents or performing more conservative therapies.
* Chronic anticoagulant therapy that could limit the safety of performing rigid therapeutic bronchoscopy in a timely manner. (I.e. Plavix within one year of drug eluding cardiac stent (DES) or 6 weeks following bare metal coronary stent)
* Unstable cardiac disease
* Allergy to silicone
* Stenting to manage vascular compression syndromes.
* Multi-drug resistant bacterial or fungal chronic infections
* Emergent/urgent clinically indicated stent.
* Chronic/permanent mechanical ventilation.
* Pure Excessive Dynamic Airway Collapse (EDAC) patients.
* Pure Pulmonary Resistance (Rp) patients.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Baseline Dyspnea Index/Transitional Dyspnea Index | Day -1
  Change in BDI/TDI over course of study
Baseline Dyspnea Index/Transitional Dyspnea Index | Day 1
  Change in BDI/TDI over course of study
Baseline Dyspnea Index/Transitional Dyspnea Index | Day 14
  Change in BDI/TDI over course of study
Baseline Dyspnea Index/Transitional Dyspnea Index | Day 30
  Change in BDI/TDI over course of study
Baseline Dyspnea Index/Transitional Dyspnea Index | Day 60
  Change in BDI/TDI over course of study
Baseline Dyspnea Index/Transitional Dyspnea Index | Day 90
  Change in BDI/TDI over course of study
Baseline Dyspnea Index/Transitional Dyspnea Index | Day 180
  Change in BDI/TDI over course of study
Ability to implant stent | Day 0
  Number of patients able to successfully receive patient-specific stent

SECONDARY OUTCOMES:
SGRQ | Day -1
  Change in Quality of Life over course of study
SGRQ | Day 60
  Change in Quality of Life over course of study
SGRQ | Day 90
  Change in Quality of Life over course of study
SGRQ | Day 180
  Change in Quality of Life over course of study
CTCAE | Day 0
  Number of adverse event(s) over course of study
CTCAE | Day 1
  Number of adverse event(s) over course of study
CTCAE | Day 14
  Number of adverse event(s) over course of study
CTCAE | Day 30
  Number of adverse event(s) over course of study
CTCAE | Day 60
  Number of adverse event(s) over course of study
CTCAE | Day 90
  Number of adverse event(s) over course of study
CTCAE | Day 180
  Number of adverse event(s) over course of study

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Pulmonary Medicine, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided
Neither the complete nor any part of the results of the study carried out under this protocol, nor any of the information provided by the sponsor for the purposes of performing the study, will be published or passed on to any third party without the consent of the study sponsor. Any investigator involved with this study is obligated to provide the sponsor with complete test results and all data derived from the study.

REFERENCES:
- [Background] Saad CP, Murthy S, Krizmanich G, Mehta AC. Self-expandable metallic airway stents and flexible bronchoscopy: long-term outcomes analysis. Chest. 2003 Nov;124(5):1993-9. doi: 10.1378/chest.124.5.1993. PMID 14605078
- [Background] Gildea TR, Downie G, Eapen G, Herth F, Jantz M, Freitag L. A prospective multicenter trial of a self-expanding hybrid stent in malignant airway obstruction. Journal of Bronchology 2008;15:221-4
- [Background] FDA public health notification: complications from metallic tracheal stents in patients with benign airway disorders. 2005. Anonymous . (, at www.fda.gov/cdrh/safety/072905-tracheal.html)
- [Background] Gershman AJ, Gildea TR, Mehta AC. Complication of metallic stent in lung transplant dehiscence. J Heart Lung Transplant. 2006 Jun;25(6):742-3. doi: 10.1016/j.healun.2006.02.008. Epub 2006 May 2. No abstract available. PMID 16730586
- [Background] Choudhary C, Bandyopadhyay D, Salman R, Gildea T, Mehta A. Broncho-vascular fistulas from self-expanding metallic stents: A retrospective case review. Ann Thorac Med. 2013 Apr;8(2):116-20. doi: 10.4103/1817-1737.109830. PMID 23741275
- [Background] Breen DP, Dutau H. On-site customization of silicone stents: towards optimal palliation of complex airway conditions. Respiration. 2009;77(4):447-53. doi: 10.1159/000205396. Epub 2009 Feb 26. PMID 19246883
- [Background] Alraiyes AH, Machuzak MS, Gildea TR. Intussusception technique of intrabronchial silicone stents: description of technique and a case report. J Bronchology Interv Pulmonol. 2013 Oct;20(4):342-4. doi: 10.1097/LBR.0000000000000009. PMID 24162120
- [Background] Tendulkar RD, Fleming PA, Reddy CA, Gildea TR, Machuzak M, Mehta AC. High-dose-rate endobronchial brachytherapy for recurrent airway obstruction from hyperplastic granulation tissue. Int J Radiat Oncol Biol Phys. 2008 Mar 1;70(3):701-6. doi: 10.1016/j.ijrobp.2007.07.2324. Epub 2007 Sep 29. PMID 17904764
- [Background] Kumar A, Alraiyes AH, Gildea TR. Amniotic Membrane Graft for Bronchial Anastomotic Dehiscence in a Lung Transplant Recipient. Ann Am Thorac Soc. 2015 Oct;12(10):1583-6. doi: 10.1513/AnnalsATS.201505-265CC. No abstract available. PMID 26448355
- [Background] Dutau H, Cavailles A, Sakr L, Badier M, Gaubert JY, Boniface S, Doddoli C, Thomas P, Reynaud-Gaubert M. A retrospective study of silicone stent placement for management of anastomotic airway complications in lung transplant recipients: short- and long-term outcomes. J Heart Lung Transplant. 2010 Jun;29(6):658-64. doi: 10.1016/j.healun.2009.12.011. Epub 2010 Feb 4. PMID 20133161
- [Background] Fortin M, MacEachern P, Hergott CA, Chee A, Dumoulin E, Tremblay A. Self-expandable metallic stents in nonmalignant large airway disease. Can Respir J. 2015 Jul-Aug;22(4):235-6. doi: 10.1155/2015/246509. PMID 26252535
- [Background] Gildea TR, Murthy SC, Sahoo D, Mason DP, Mehta AC. Performance of a self-expanding silicone stent in palliation of benign airway conditions. Chest. 2006 Nov;130(5):1419-23. doi: 10.1378/chest.130.5.1419. PMID 17099019